CLINICAL TRIAL: NCT07257991
Title: Comparison of Dressing Materials of Donor Site of Split-thickness Skin Graft; Paraffin Mesh Gauze vs Povidone-Iodine Foam at SMBB Institute of Trauma Karachi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Mohtarma Benazir Bhutto Institue of Trauma (Other)
Responsible Party: Principal Investigator, Saba Asif, Postgraduate Trainee, Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB000195/SMBBIT/Approval/2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Skin Graft Wounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG GROUP (Active Comparator): Paraffin gauze dressing will be used.
  Interventions: Procedure: Paraffin mesh gauze dressing for donor site of Split-thickness skin graft
- PI GROUP (Experimental): Povidone-iodine foam dressing will be used in this group.
  Interventions: Procedure: Povidine-iodine foam dressing for donor site of Split-thickness skin graft

INTERVENTIONS:
Procedure: Povidine-iodine foam dressing for donor site of Split-thickness skin graft — A sterile, medical-grade open-cell polyurethane foam will be cut to fit the split-thickness skin graft donor site and soaked in 3% povidone-iodine solution immediately before application. The foam dressing will be applied to the donor site under aseptic conditions and secured with a sterile secondary dressing of gauze and crepe bandage.
  The initial dressing will be left undisturbed for 7 days unless early change is required due to bleeding, leakage, loosening, or signs of infection. The donor site will first be assessed on day 7, and subsequently every alternate day until complete re-epithelialization. At each assessment, the dressing will be changed only if clinically indicated.
  Arms: PI GROUP
Procedure: Paraffin mesh gauze dressing for donor site of Split-thickness skin graft — A sterile paraffin-impregnated mesh gauze dressing will be applied directly over the donor site under aseptic conditions. The dressing will be covered with sterile secondary gauze and secured with crepe bandage. The initial dressing will be left undisturbed for 7 days unless early change is required for bleeding, leakage, or infection. The donor site will be assessed on day 7 and every alternate day thereafter until complete re-epithelialization, and the dressing will be changed only if clinically indicated.
  Arms: PG GROUP

SUMMARY:
The goal of this clinical trial is to learn if povidone-iodine foam dressing is better in achieving complete reepithelialization of donor site wounds after harvest of split-thickness skin graft as paraffin mesh gauze.

The main questions it aims to answer are:

Does povidone-iodine foam dressing promotes complete reepithelialization earlier in comparison? Which type of dressing will require fewer replacements? Which type of dressing material is associated with less pain?

Non-probability consecutive sampling method will be used and participants divided in two groups. Donor site wounds after split-thickness skin graft harvest will be dressed using two different dressing materials. Participants will be followed until complete epithelialization with change of dressing on follow-ups if required. Complete epithelialization is usually achieved within two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing skin graft with donor site size between 25 to 200 cm2

Exclusion Criteria:'

* Patients wit history of disease impairing wound healing (Diabetes, Malignancy, Cancer, taking immunosuppressants)
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete reepithelialization at day 14 | From the day of procedure till complete reepithelialization, nearly 14 days
  Measurement name is percentage of patients. Measurement tool will be clinical observation/ visual assessment by principal investigator defined as 100% wound healing.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pak CS, Park DH, Oh TS, Lee WJ, Jun YJ, Lee KA, Oh KS, Kwak KH, Rhie JW. Comparison of the efficacy and safety of povidone-iodine foam dressing (Betafoam), hydrocellular foam dressing (Allevyn), and petrolatum gauze for split-thickness skin graft donor site dressing. Int Wound J. 2019 Apr;16(2):379-386. doi: 10.1111/iwj.13043. Epub 2018 Nov 26. PMID 30479060
- See also: Comparison of the efficacy and safety of povidone-iodine foam dressing (Betafoam), hydrocellular foam dressing (Allevyn), and petrolatum gauze for split-thickness skin graft donor site dressing — https://pubmed.ncbi.nlm.nih.gov/30479060/